CLINICAL TRIAL: NCT02275741
Title: Study to Investigate the Immune Response and Safety of Prophylactic Vaccines in Patients Treated for Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Dr. med. Micha Loebermann (Other)
Responsible Party: Sponsor-Investigator, Dr. med. Micha Loebermann, Deputy Head, Department of Tropical Medicine an Infectious Diseases, University of Rostock
Organization: University of Rostock (Other)
Other Study IDs: UMR-MS2012
Record Dates: First submitted 2014-10-22; First posted 2014-10-27 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Vaccine; Antibody response; relaps rate; expanded disability status scale
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Tetanus Toxoid; Influenza Vaccines; Hepatitis A Vaccines; Hepatitis B Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum sample
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: prophylactic vaccine (tetanus, diphtheria, pertussis, poliomyelitis, influenza, hepatitis A, hepatitis B, tick-borne encephalitis, meningococcal, pneumococcal) — Publically recommended protective vaccines in MS patients, vaccination applied according to the manufacturers description

SUMMARY:
The aim of this study is to determine whether prophylactic vaccines recommended are effective and safe in patients with multiple sclerosis(MS) under MS-specific therapy.

DETAILED DESCRIPTION:
Protective vaccines against communicable diseases are of major importance in patients with autoimmune diseases or impaired immune response. In patients with multiple sclerosis bacterial or viral infections may lead to disease progression and vaccines can protect from these infections and prevent disease progression. Fear of possible side effects of vaccines have led to a general restraint regarding vaccination of patients with MS. However, previous studies have not shown an increased risk of disease progression following Hepatitis B vaccination and even a reduced progression rate in relapsing-remitting MS after tetanus/diphtheria vaccination.

Various disease modifying treatments (DMT) are available for MS, most of these therapies lead to an impairment of the immune system affecting the immune response to vaccination. Additionally, live attenuated vaccines may lead to severe side-effects if used in patients under DMT treatment. Testing immune response after vaccination may be prudent in subjects undergoing DMT to assure vaccination success since only a limited number of studies have investigated immune response after vaccination in patients with MS undergoing DMT.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of Multiple Sclerosis
* Age: 18 - 70 years
* Indication for vaccination (according to public recommendation)
* Written informed consent

Exclusion Criteria:

* Current relapse of MS
* Unstable disease
* Contraindication for vaccination (acute infection, fever, allergy to vaccine)
* Unable to comply with study procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: relapsing remitting multiple sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2009-10; Primary Completion 2015-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Specific antibody response to vaccination | four weeks
  Serum samples are evaluated before and 4 Weeks after vaccination

SECONDARY OUTCOMES:
MS relapse rate | 12 months
  Course of MS is evaluated by relapse rate and EDSS (expanded disability status scale) is evaluated prior to and at month 6 and 12 after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Uwe K Zettl, Prof. Dr., Principal Investigator — University of Rostock
Locations (1):
- University of Rostock, Rostock, Germany

REFERENCES:
- [Result] Metze C, Winkelmann A, Loebermann M, Hecker M, Schweiger B, Reisinger EC, Zettl UK. Immunogenicity and predictors of response to a single dose trivalent seasonal influenza vaccine in multiple sclerosis patients receiving disease-modifying therapies. CNS Neurosci Ther. 2019 Feb;25(2):245-254. doi: 10.1111/cns.13034. Epub 2018 Jul 25. PMID 30044050
- [Derived] Winkelmann A, Metze C, Frimmel S, Reisinger EC, Zettl UK, Loebermann M. Tick-borne encephalitis vaccination in multiple sclerosis: A prospective, multicenter study. Neurol Neuroimmunol Neuroinflamm. 2020 Jan 9;7(2):e664. doi: 10.1212/NXI.0000000000000664. Print 2020 Jan. PMID 31919278